CLINICAL TRIAL: NCT04188327
Title: Utility of Early Serial Stellate Ganglion Block in Acute Herpes Zoster of Face and Neck
Brief Title: Stellate Ganglion Block in Herpes Zoster
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Collaborators: Mohamad Gamal Elmawy, M.D (Unknown)
Responsible Party: Principal Investigator, Sameh Abdelkhalik Ahmed Ismaiel, Dr, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 33426/10/10
Record Dates: First submitted 2019-11-28; First posted 2019-12-05 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Pain; Neuropathic
Keywords: Herpes Zoster; Stellate ganglion; Post-herpetic neuralgia
MeSH Terms: conditions — Pain; Herpes Zoster; Neuralgia, Postherpetic

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: * The patients will be blind through the use of closed sealed envelops.
  * The investigator will be blind through the use of sham block in the control group.
  * The measurement will be collected by anesthesiologist not participating in the study and blinded to its group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group(Group I) (Sham Comparator): Patients will receive sham stellate ganglion block weekly for three times
  Interventions: Procedure: Sham Stellate ganglion block
- Stellate Ganglion block group (Group II) (Experimental): Patients will receive stellate ganglion block weekly for three times with injection of 6ml bupivicain 0.25%+ 1 ml methylpredinosolone 40mg
  Interventions: Procedure: Stellate ganglion block

INTERVENTIONS:
Procedure: Stellate ganglion block — While the patient is in a supine position with slight neck extension and rotation to the contralateral side, in-plane ultrasound guided stellate ganglion block will be performed with injection of 7 ml injectate (6ml bupivicain 0.25%+ 1 ml methylpredinosolone 40mg).
  Each patient will receive:
  * Acyclovir 800 mg orally every 5 times per day 7 days.
  * Pregabalin start with 50 mg orally every 8hours for 7 days then increase to 150 mg every 12 hours
  Arms: Stellate Ganglion block group (Group II)
Procedure: Sham Stellate ganglion block — The patient will be positioned supine with slight neck extension and rotation to the contralateral side. Under US guidance, a sham stellate ganglion block will be performed with injection of a 1ml injectate of normal saline will be done while observing the dissection between the carotid artery and the longus colli muscle.
  Each patient will receive:
  * Acyclovir 800 mg orally every 5 times per day for 7 days.
  * Pregabalin start with 50 mg orally every 8hours for 7 days then increase to 150 mg every 12 hours
  Arms: Control group(Group I)

SUMMARY:
Patient who will be presented to Tanta University Hospitals complaining of acute herpes zoster with onset of vesicular eruption less than 7 days will be included in this clinical study.

Patients will be excluded if they refused participation, had allergy to local anesthetics, coagulopathy, local infection, glaucoma, or neurological deficit.

All the patients will receive acyclovir (antiviral therapy) and pregablin (analgesic) and the patients will be classified into two groups:- Group I (control group): Patients will receive sham block weekly for three times Group III (SGB group): Patients will receive stellate ganglion block weekly for three times

The time of first block after the onset of vesicular eruption, the incidence of PHN, NPRS at visit, duration of acute HZ , duration of PHN (if occurred), and the incidence of complication will be measured.

DETAILED DESCRIPTION:
This prospective randomized study will be carried out on adult patients complaining of acute herpes zoster presented at Tanta University Hospitals after approval from ethics committee for twelve months.

An informed consent will be taken from each patient. All data of patients will be confidential with secret codes and private file for each patient. All given data will be used for the current medical research only.

Any unexpected risk encountered during the course of the research will be cleared to the participant as well as to the Ethical Committee on time. Every patient will receive an explanation to the purpose of the study and will have a secret code number to ensure privacy of the participants and confidentiality of their data.

The study will be terminated in case of incidence of severe hypotension no responding to ephedrine (Mean arterial blood pressure less than 60 mmHg) or severe bradycardia not responding to atropine (Heart rate less than 40 b/min). The participants and the ethical committee will be announced.

There will be adequate supervision to maintain the privacy of patients and confidentiality of data. There will be no conflict of interest, nor conflict with religion, law, or society standards. The research will be beneficial to the society and has no risk of environmental pollution.

After inclusion, adequate history taking, clinical examination, and laboratory investigation (as needed) will be done for all patients. Every patient will be educated about the use of the 0-10 numerical rating scale for pain assessment (NPRS: with endpoints of 'no pain' and 'worst pain').

Each patient will receive:

* Acyclovir 800 mg orally every 5 times per day (for immuno-compromised patients 10 mg/kg IV 3 times per day) for 7 days.
* Pregabalin start with 50 mg orally every 8hours for 7 days then increase to 150 mg every 12 hours

Groups:

Participants will be divided into two groups; each group consists of (88) patients. The sample size calculation was made using Epi-Info software program created by the WHO

* Group I (control group): Patients will receive sham block weekly for three times
* Group II (SGB group): Patients will receive stellate ganglion block weekly for three times

Equipment

* 10-mL syringe - For local anesthetic
* 22- or 25-gauge, 1.5-inch short-bevel needle
* Skin temperature monitor
* Ultrasound machine with a 6-12 MHz linear type probe.
* Appropriate equipment and medications for medical resuscitation

Technique of SGB:

The patient will be positioned supine with slight neck extension and rotation to the contralateral side. After adequate asepsis of the neck, the probe will be placed perpendicular to tracheal axis at the cricoid cartilage. An initial scan will be obtained to identify structures: thyroid gland, carotid artery and jugular vein.

The transverse process at C6 should be identified as the initial landmark because of its prominent anterior tubercle (The Chassaignac tubercle). The long muscle of the neck (longus colli) is found above it.

The puncture should be in-plane to see the tip of the needle all the time. The needle will be directed medially until it passes through the deep cervical fascia above the longus colli muscle.

Considering repeated aspiration test, a 7 ml injectate (for SGB group: 6ml bupivicain 0.25%+ 1 ml methylpredinosolone 40mg) will be done while observing the dissection between the carotid artery and the longus colli muscle.

After finishing the block:

The patient will be transferred to the recovery room for 30-60 min to assess any potential complications. After that he will be discharged.

Review appointments will be arranged weekly for 4 weeks then every 2 weeks for 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who is presented to the pain clinic, diagnosed with acute herpes zoster of the face and/ or neck with onset of vesicular eruption less than seven days

Exclusion Criteria:

* Patient refusal or un-cooperation
* Known history of allergy to local anesthetics
* Local infection at the site of the block
* Platelet count less than 75,000/ cc
* Neurological deficit in the upper limb
* Glaucoma
* Bradycardia

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2025-02-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Post-herpetic neuralgia | within 3 months of the last stellate ganglion block
  The incidence of chronic neuropathic pain in the face or the neck after herpes zoster

SECONDARY OUTCOMES:
The duration of herpes zoster | Through study completion, an average of 1 year
  The time from diagnosis of HZ till resolving of it

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Ismaiel, M.D, Principal Investigator — Lecturer of Anesthesia and Intensive Care, Tanta University
Locations (3):
- Egypt (3):
  - Faculty of Medicine, Tanta, Algharbia
  - Faculty of Medicine, Al Fayyum
  - Tanta University hospitals, Tanta

IPD SHARING:
Plan to Share IPD: No
Once the study had been successfully completed, the data will be shared for other researchers.